CLINICAL TRIAL: NCT02385175
Title: The Accuracy of Tests of Eustachian Tube Function
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, James Tysome, Principle Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 166405
Record Dates: First submitted 2015-03-03; First posted 2015-03-11 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Eustachian Tube Dysfunction
Keywords: Eustachian tube; test accuracy; clinical test; questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with suspected Eustachian tube dysfunction: Age 18+ with possible Eustachian tube dysfunction on the basis of symptoms and examination findings.
  Interventions: Other: Different objective clinical tests of Eustachian tube function; Other: Different patient-completed questionnaires relating to Eustachian tube dysfunction

INTERVENTIONS:
Other: Different objective clinical tests of Eustachian tube function
Other: Different patient-completed questionnaires relating to Eustachian tube dysfunction

SUMMARY:
The Eustachian tube links the middle ear to the back of the nose and is designed to open to allow the pressure in the air-filled middle ear to be equal to external (atmospheric) pressure. In some people this system fails to work properly leading to abnormal pressure in the middle ear, and complications such as middle ear fluid ('glue ear') or damage to the ear drum. The abnormal function of the Eustachian tube is called 'Eustachian tube dysfunction'. An affected person may feel pressure, pain or other symptoms in their ear, and their hearing can be temporarily or permanently reduced.

This study is designed to find out which of a number of simple tests is best at detecting if the Eustachian tube is performing normally. Both patient-completed questionnaires and clinical tests using specialist machines will be compared as a way of diagnosing Eustachian tube dysfunction.

A group of adults aged 18 and above, and children aged 5-17 years with normal ears, and a similar group of people that are already known to have Eustachian tube dysfunction, will both take six different tests and complete four different questionnaires. The differences in the results between the group with ETD and the healthy group will be compared. The results for each test or questionnaire will be compared to see which is best at telling the healthy and Eustachian tube function groups apart, and therefore at diagnosing Eustachian tube dysfunction. The investigators will also look to see if a combination of one or more of the tests or questionnaires is best at diagnosing the disease.

The results of this study hope to provide a test or combination of tests that can be used on a daily basis by ENT doctors. The assessment technique would also be helpful in researching and comparing new treatments for ETD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with Eustachian tube dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Test sensitivity and specificity for assignment of patients to case or control groups | Patients will undertake each assessment once in a single session
  Each test will be interpreted as per standard practice, using a validated method where available

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom